CLINICAL TRIAL: NCT05257525
Title: Impact of Chest Wall Mechanics on Lung and Cardiovascular Function During Delayed Sternal Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Luciana Rodriguez Guerineau, Staff Physician, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1000075860
Record Dates: First submitted 2022-01-25; First posted 2022-02-25 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Palliation of Congenital Heart Diseases; Cardiopulmonary Bypass; Chest Wall Mechanics; Neonatal Delayed Sternal Closure
Keywords: chest wall mechanics; congenital heart disease; neonates; delayed sternal closure; cardiopulmonary bypass
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Tidal Volume

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Univentricular physiology (Other): Neonates with univentricular physiology
  Interventions: Other: Esophageal manometry catheter at various PEEP levels and tidal volumes
- Biventricular physiology (Other): Neonates with biventricular physiology
  Interventions: Other: Esophageal manometry catheter at various PEEP levels and tidal volumes

INTERVENTIONS:
Other: Esophageal manometry catheter at various PEEP levels and tidal volumes — Participants will undergo placement of an esophageal manometry catheter before planned sternal closure. This catheter will be used to measure esophageal pressure which is a surrogate for pleural (intrathoracic) pressure. Esophageal pressure will then be used to estimate changes in respiratory system mechanics and hemodynamics following sternal closure and across different levels of positive end-expiratory pressure (PEEP) and tidal volumes.

SUMMARY:
This study aims to describe chest wall mechanics during delayed sternal closure (DSC) in neonates following cardiopulmonary bypass or palliation of congenital heart diseases.

DETAILED DESCRIPTION:
This research study is being done so that investigators can understand the complex interactions between the heart, the lungs and the chest wall after heart surgery. Understanding this may guide future care that can help patients with their recovery from heart surgery.

The heart and lungs work together to make sure the body has the oxygen-rich blood it needs to function properly. The chest wall protects the heart, lungs, and other important organs. Investigators would like to learn how a patient's chest wall contributes to the heart and lungs interaction when the chest is left open after heart surgery.

Investigators will be using a device called an esophageal pressure catheter to estimate the pressure that is transmitted to the lungs and heart, called pleural pressure. Previous research has shown that this pressure measurement is used to adjust the breathing machine for patients with lung diseases. Measuring the pressure transmitted to the lungs and heart after heart surgery and delayed chest wall closure may help investigators understand how the chest wall contributes to the heart and lung interaction.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent provided by parent or primary guardian.
2. Aged <28 days of life at the time of cardiac surgery.
3. Undergone surgery using CPB for congenital heart disease.
4. Undergoing DSC in CCCU.

Exclusion Criteria:

1. Gestational age < 37 weeks or weight < 2 kg at the time of surgery.
2. Endotracheal tube leak >20%.
3. Need of extracorporeal support (ECMO), inhaled nitric oxide.
4. Pre-existing pulmonary disease (For example: Congenital diaphragmatic hernia).
5. Pre-existing or new arrhythmia that can impact hemodynamic assessment.
6. Severe coagulopathy or any other contraindication for the insertion of a nasogastric catheter (e.g., history of tracheo-esophageal fistula).

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with successful insertion and measurement of esophageal pressures | Immediately prior to chest closure and repeated measurements after chest closure
  Investigators hypothesize that successful esophageal catheter placement and measurement of Pes (full data set) will occur in ≥80% of enrolled subjects.

SECONDARY OUTCOMES:
End-inspiratory and end-expiratory transpulmonary pressure | Prior to and immediately after sternal chest wall closure procedure
  cmH20
Transmural systolic pressures | Prior to and immediately after sternal chest wall closure procedure
  mmHg
Transmural diastolic pressures | Prior to and immediately after sternal chest wall closure procedure
  mmHg
Chest wall and lung compliance | Prior to and immediately after sternal chest wall closure procedure
  mL/cmH20
Changes in transmural pressures | Prior to and immediately after sternal chest wall closure procedure
  mmHg
Duration of inotropic support | At 30 days post-operation or discharge (whichever comes first)
  Hours
Duration of support with supplemental oxygen | At 30 days post-operation or discharge (whichever comes first)
  Days
Length ICU Stay | At 30 days post-operation or discharge (whichever comes first)
  Days
Duration of mechanical ventilation | At 30 days post-operation or discharge (whichever comes first)
  Hours
Length of Hospital Stay | At 30 days post-operation or discharge (whichever comes first)
  Days
Mortality | At 30 days post-operation or discharge (whichever comes first)
  Yes/No

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Rodriguez Guerineau, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All de-identified individual participant data (IPD) that underlie results in a publication will be shared upon request. The study protocol, statistical analysis plan, informed consent form, and analytic code will be shared starting (6 months after publication or starting January 2023, whichever comes first) upon request in writing.
  Requests for IPD will be reviewed by the study PI and SickKids institute. IPD will be provided to researchers interested in furthering academia and research development only. IPD requests may also be subjected to SickKids' institutional agreements/contracts. IPD mechanism of sharing and types of analysis/data shared will be directed and determined by SickKids' institutional research contracts requirements.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 6 months after publication or starting January 2023, whichever comes first
Access Criteria: Requests for IPD will be reviewed by the study PI and SickKids institute. IPD will be provided to researchers interested in furthering academia and research development only. IPD requests may also be subjected to SickKids' institutional agreements/contracts. IPD mechanism of sharing and types of analysis/data shared will be directed and determined by SickKids' institutional research contracts requirements.